CLINICAL TRIAL: NCT05133154
Title: LIQUID BIOPSY IN Low-grade Glioma Patients
Acronym: GLIOLIPSY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RECHMPL20_0671; 2021-A00584-37 (Other: ANSM)
Record Dates: First submitted 2021-10-25; First posted 2021-11-24 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Glioma
Keywords: Low-grade glioma; High-grade glioma; Circulating tumor cells; Circulating biomarker; Tumor-educated platelets
MeSH Terms: conditions — Glioma; Neoplastic Cells, Circulating | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: The subjects will be included in the 3 following groups :
  * Group 1 : "Low-grade glioma" group: n=30
  * Group 2 : "High-grade glioma" group: n=10
  * Group 3 : "Control" (patients undergoing brain surgery for a non-tumor disease) group: n=10
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Patients with low-grade glioma (Other): Group 1
  Interventions: Biological: Blood samples
- Patients with high-grade glioma (Other): Group 2
  Interventions: Biological: Blood samples
- Patients undergoing brain surgery for a non-tumor disease (Other): Group 3
  Interventions: Biological: Blood samples

INTERVENTIONS:
Biological: Blood samples — In total, about 20 ml of blood will be collected on EDTA tubes : collection of CTCs, TEPs and biobanking (V0, V1 and V2)

SUMMARY:
Diffuse low-grade gliomas (DLGG) (or WHO grade II gliomas) are rare tumors, with an incidence estimated at 1/105 person-year. DLGG are characterized by a continuous growth and an unavoidable anaplastic transformation. DLGG malignant progression is classically characterized by a continuum, from grade II to grade III or IV tumors.

To date, the histomolecular diagnosis of lower grade gliomas (that is, grade II and III gliomas) is achieved on tumor samples obtained from surgical resection or biopsy. Indeed, whereas brain MRI is often suggestive of DLGG, there is a need for a histological confirmation of diagnosis prior to any medical treatment. Moreover, MRI features to not always accurately predict the tumor grade, with grade II tumor presenting with contrast enhancement or non-enhancing authentic grade III tumors.

In this setting, the value of liquid biopsy (in blood or cerebrospinal fluid CSF) as a non-invasive, disease-associated biomarker has gained interest in the past decade, either at tumor diagnosis or to monitor tumor evolution in order to guide patient management and to detect changes of molecular features over time. While extracranial metastasis of glioma rarely occurs, recent reports suggest the possible presence of circulating tumor cells (CTCs) in blood of high-grade glioma patients. Beside CTCs, other circulating biomarkers have been recently investigated in glioma, including circulating tumor DNA, microRNA or tumor-educated platelet (TEP) RNA. Some of these techniques allow genome-wide characterization of RNA/DNA contents.

However, these studies are all small exploratory studies that have mainly included glioblastoma (grade IV glioma) patients rather than lower-grade gliomas, or glioma patients with no precision on tumor grade. Moreover, some of these studies analyzed samples performed after the patient received a medical oncological treatment (chemotherapy or radiation therapy). They advocate for the search of a circulating signature that would not be restricted to biomarkers directly derived from the tumor but include markers induced at a distance by the tumor. Indeed, slow-growing DLGG are likely to induce a systemic reaction to allow, for many years, an immuno-tolerance of the tumor. This reaction could have an impact on peripheral blood cells, including their RNA content.

In this study, the investigators aim at conducting an exploratory study in DLGG patients to explore the value of several blood-based biomarkers for the disease diagnosis and/or monitoring.

DETAILED DESCRIPTION:
This study is a prospective, exploratory and bi-centric study.

The primary objective is to evaluate the presence of CTCs in a preoperative sample for the 3 following groups : patients with low-grade glioma, patients with high-grade glioma and patients undergoing neurosurgery for a non-tumor disease.

Visits in this study are as follows :

Inclusion Visit (V0) : 2 days (+/- 2 days) before brain surgery

Postoperative visits :

* Visit 1: 2 days (+/- 2 days) following brain surgery
* Visit 2: 3 months (+/- 1 month) following brain surgery

ELIGIBILITY:
Inclusion Criteria:

* Adult patient aged ≥ 18, no age limit
* A signed informed consent obtained before any study specific procedures
* Patient affiliated to a French social security system
* Patient ability to understand experimental procedures
* Patient able to speak, read and understand French

Also for the "Low-grade glioma" group, the following inclusion criteria applies:

- Brain surgery for a suspected low-grade tumor, histologically confirmed on tumor sample

Also for the "High-grade glioma" group, the following inclusion criteria applies:

- Brain surgery for a suspected high-grade glioma, histologically confirmed on tumor sample

Also for the "Control group, the following inclusion criteria applies:

- Brain surgery for a non-tumor disease (cavernoma, arteriovenous malformation)

Exclusion Criteria:

* Legal incapacity or physical, psychological social or geographical status interfering with the patient's ability to sign the informed consent or to terminate the study
* Pregnant and/or breastfeeding women (this will be checked in declarative way)
* Patients with medical history of cancer other than the brain tumor, whatever the treatment received

Also, for the "Low-grade glioma" group, the following exclusion criteria applies:

* Previous chemotherapy or radiation therapy for the low-grade glioma (but previous surgery/ies is/are allowed)
* No indication for chemotherapy for 6 month after surgery

Also, for the "High-grade glioma" group, the following exclusion criteria applies:

- Previous chemotherapy or radiation therapy for the glioma

Also, for the "control" group, the following exclusion criteria applies:

- Diagnosis or suspicion of primary or secondary brain tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with CTCs (>0) in a preoperative sample for the 3 following groups (patients with low-grade glioma, patients with high-grade glioma and patients undergoing neurosurgery for a non-tumor disease) | 14 months

SECONDARY OUTCOMES:
Number and characteristics of CTCs (in patients with CTCs) in a preoperative sample for the 3 groups of patients | Baseline
Platelets RNA profile in a preoperative sample for the 3 groups | Baseline
Number, characteristics of CTCs (in patients with CTCs) and platelets profile in a postoperative sample for the 3 groups | 2 days following brain surgery
Number, characteristics of CTCs (in patients with CTCs) and platelets profile in a postoperative sample for the 3 groups | 3 months following brain surgery
FLAIR tumor volume | Baseline
  calculated by manual segmentation of the tumor borders on preoperative T2/FLAIR weighted MRI
Spontaneous growth speed | Baseline
  calculated as the evolution in mm/year of the mean tumor diameter derived from tumor volume (mm/year)
Contrast enhancement | Baseline
  defined on post Gadolinium pre-operative MRI (presence or absence)
Tumor location | Baseline
ECOG performance status | Baseline + 3 months following brain surgery
Tumor-associated symptoms | Baseline + 3 months following brain surgery
Time interval since the first symptoms and the first MRI | Baseline
Associated drugs (antiepileptic drugs, corticosteroids) | Baseline + 3 months following brain surgery
Previous treatments for the tumor | Baseline + 3 months following brain surgery
WHO classification | 3 months following brain surgery
IDH status | 3 months following brain surgery
1p19q status | 3 months following brain surgery
ATRX status | 3 months following brain surgery
Proliferation index (Ki67) | 3 months following brain surgery
Presence of foci of malignant transformation | 3 months following brain surgery

CONTACTS AND LOCATIONS:
Overall Officials: Catherine PANABIERES, MCU-PH, Ph.D., Study Director — University Hospital, Montpellier
Locations (1):
- University Hospital, Montpellier, Montpellier, France